CLINICAL TRIAL: NCT04964661
Title: Incidence of Sacro-iliac (SI) Joint Anomalies on MRI: Differentiation Criteria in Women With Spondyloarthritis (SpA
Brief Title: Incidence of MRI Sacro-Iliac (SI) Joint Anomalies in Women With Spondyloarthritis (SpA)
Acronym: MISIA 2
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0612
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Spondylarthritis
Keywords: Diagnostic Imaging; Magnetic Resonance Imaging; Sacroiliac Joint anomalies
MeSH Terms: conditions — Spondylarthritis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SpA women MRI: Women affected by spondyloarthritis and performed a sacroiliac MRI
  Interventions: Other: Medical Imaging

INTERVENTIONS:
Other: Medical Imaging — MRI imaging

SUMMARY:
Retrospective study comparing the incidence of inflammatory and structural lesions seen on MRI of the sacro-iliac (SI) joints in a population of women affected by spondyloarthritis (SpA) and control women population (MISIA study NCT02956824).

A previous study (MISIA) demonstrate SpA may be misdiagnosed on MRI in postpartum women due to increased stress on the joint following pregnancy and childbirth, as MRI of the SI joints may show lesions that could mimics SpA.

The primary objective of this study is to compare the incidence and pattern of MRI inflammatory and structural lesions of the SI joints between SpA and control women, and determine differentiation criteria in SpA women.

ELIGIBILITY:
Inclusion criteria:

* Women aged 18 to 50 years old
* SpA diagnosed
* Pelvis MRI performed

Exclusion criteria:

- Pelvis MRI unavailable

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18 to 50 years old Affected by spondyloarthritis Performed sacroiliac joint MRI
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of MRI inflammatory of the sacroiliac joints | day 1
  MRI inflammatory of the sacroiliac joints in the population of women affected by SpA

SECONDARY OUTCOMES:
Rate of structural lesions of the sacroiliac joints | day 1
  structural lesions of the sacroiliac joints in the population of women affected by SpA

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CYTEVAL, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC